CLINICAL TRIAL: NCT04202809
Title: Prospective Phase-II Trial of Induction Chemotherapy and Chemoradiotherapy Plus/Minus the PD-L1 Antibody Durvalumab Followed by Surgery or Definitive Chemoradiation Boost and Consolidation Durvalumab in Resectable Stage III NSCLC.
Brief Title: Phase-II Trial of Induction Chemotherapy and Chemoradiotherapy Plus/Minus Durvalumab and Consolidation Immunotherapy in Patients With Resectable Stage III NSCLC.
Acronym: ESPADURVA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Essen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESPADURVA
Record Dates: First submitted 2019-12-04; First posted 2019-12-18 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: NSCLC, Stage III
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chemo- and Radiochemotherapy + Durvalumab (Experimental)
  Interventions: Drug: Durvalumab
- Chemo- and Radiochemotherapy (No Intervention)

INTERVENTIONS:
Drug: Durvalumab — Durvalumab is given earlier as registered, during chemotherapy and radiotherapy in treatment Arm A
  Arms: Chemo- and Radiochemotherapy + Durvalumab

SUMMARY:
To compare a complex induction multimodality protocol (ESPATUE) + concurrent immunotherapy with PD-L1 antibody Durvalumab given every three weeks to the same induction multimodality protocol without Durvalumab immunotherapy induction followed by definitive local treatment (surgery for those considered resectable or chemoradiation boost for those not considered to be R0-resectable) followed by consolidation Durvalumab treatment in both arms.

ELIGIBILITY:
Inclusion Criteria:

1. Body weight >30 kg
2. Age ≥ 18 years and < 75 years
3. Male or female patients. Female (as well as male) patients have to take care of effective measures of anticonception
4. Histologically proven non-small cell lung cancer
5. Selected patients with non-small cell lung cancer stages IIIA and IIIB:
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
7. Resectable disease at the time of inclusion
8. Fulfillment of adequate criteria for functional and medical resectability as described in the European Respiratory Society (ERS)/European Society of Thoracic Surgeons (ESTS) guidelines [Brunelli et al 2009] and acceptable general clinical condition for multimodality treatment (interdisciplinary committee)
9. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. Written informed consent and any locally required authorization (e.g, European Union [EU] Data Privacy Directive in the EU) obtained from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluations.
10. Must have a life expectancy of > 12 weeks
11. Adequate normal organ and marrow function
12. Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:
13. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
14. Stable cardiac function (no Myocardial infarction (MI) within 6 months, no heart failure according to New York Heart Association (NYHA) III-IV).

Exclusion Criteria:

1. resectable IIB or selected IIIA (T3N0; T3N1)
2. unresectable disease pre-treatment
3. mixed histology with areas of small cell carcinoma (neuroendocrine markers)
4. clinically symptomatic vena cava superior syndrome
5. diffuse mediastinal involvement
6. patients with T3N3 and T4N3 tumors (IIIC according to International Association for the Study of Lung Cancer (IASLC)/Union Internationale Contre le Cancer (UICC) 8)
7. invasion of the thoracic aorta (T4 - aorta)
8. invasion of the heart (except left atrium - T4 - heart)
9. invasion of the esophagus (T4 - esophagus)
10. invasion of spine (T4 - spine)
11. (full blown) Pancoast-syndrome in tumors of the superior sulcus (T3-4 Nx)
12. malignant (positive) pericardial effusion (M1a - pericardial effusion)
13. malignant (positive) pleural effusion (M1a - pleural effusion)
14. involvement of the contralateral hilar nodes (if any data available)
15. endobronchial tumor extension to the contralateral main stem bronchus
16. ipsi- or contralateral supraclavicular nodes (N3 - supraclavicular nodes)
17. lung or heart function not allowing at the time of inclusion the intended surgical procedure
18. previous administration of chemotherapy and/or radiotherapy
19. previous immunotherapy
20. insufficient patients compliance (e.g. symptomatic psychiatric disorder)
21. loss of weight > 10 % in the last six months
22. missing written informed consent or definitive refusal for participation
23. Participation in another clinical study with an investigational product during the last 12 months
24. Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study
25. Must not have required the use of additional immunosuppression other than corticosteroids for the management of an Adverse Event (AE), not have experienced recurrence of an AE if re-challenged, and not currently require maintenance doses of > 10 mg prednisone or equivalent per day
26. History of idiopathic pulmonary fibrosis, pneumonitis (including drug induced), organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia, etc.), or evidence of active pneumonitis on screening chest CT scan
27. Any concurrent chemotherapy, Intraperitoneal (IP), biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.
28. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IP. Note: Local surgery of isolated lesions for palliative intent is acceptable.
29. History of allogenic organ transplantation.
30. History of a stem cell transplantation
31. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.]).
32. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent
33. History of another primary malignancy
34. History of active primary immunodeficiency
35. Active infection including tuberculosis (TB) (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive Hepatitis B Virus (HBV) surface antigen (HBsAg) result), hepatitis C, or human immunodeficiency virus (positive HIV ½ antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody (anti-HBc) and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
36. Current or prior use of immunosuppressive medication within 14 days before the first dose of Durvalumab.
37. Current or prior use of immunostimulatory agents within 14 days before the first dose of Durvalumab.
38. Receipt of live attenuated vaccine within 90 days prior to the first dose of IP. Note: Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 90 days after the last dose of IP.
39. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of Durvalumab monotherapy.
40. Known allergy or hypersensitivity to Durvalumab or any excipient

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-01-13 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 2 years
  Two-year progression-free survival rate

SECONDARY OUTCOMES:
Overall survival | after 1, 2, 3, 4 and 5 years
2-y-overall survival rate | 2 years
Functional response | Week 15
  to investigate functional response (PET-CT-scan) to induction therapy prior to thoracotomy
RECIST response (induction) | Week 9
  to investigate RECIST response to induction therapy in the whole Population and in both arms.
RECIST criteria | Through study completion, an average of every 2 months for up to 11 months
  Radiological response
EORTC QLQ-C30 | Through study completion, an average of every 6 weeks for up to 11 months
  Quality of life (QLQ-C30)
EORTC QLQ-LC13 | Through study completion, an average of every 6 weeks for up to 11 months
  Quality of life (QLQ-Lung Cancer 13(LC13))
FACT-L | Through study completion, an average of every 6 weeks for up to 11 months
  Quality of life (Functional Assessment of Cancer Therapy-Lung (FACT-L))

CONTACTS AND LOCATIONS:
Overall Officials: Wilfried Eberhardt, PD MD, Principal Investigator — University Hospital, Essen
Locations (7):
- Germany (7):
  - Klinikum rechts der Isar - Technische Universität München, Munich, Bavaria
  - Universitätsklinikum Essen, Essen
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Lungenklinik Hemer Deutscher Gemeinschafts-Diakonieverband GmbH, Hemer
  - Pius-Hospital Oldenburg, Oldenburg
  - Universitätsklinikum Regensburg, Regensburg
  - Robert-Bosch-Krankenhaus, Stuttgart

IPD SHARING:
Plan to Share IPD: No